CLINICAL TRIAL: NCT03003507
Title: Glycemic Index Variation During Low-carbohydrate Enteral Formula With and Without Fructose in Critically Ill Patients: A Cross-over Randomized Clinical Trial
Brief Title: Glycemic Index Variation During Low-carbohydrate Enteral Formula With and Without Fructose in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Principal Investigator, Magali Kumbier, Nutritionist, Hospital Moinhos de Vento
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: v4n3n8xw
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Critical Illness
Keywords: Hyperglycemia; Fructose; Diabetes mellitus; Enteral Nutrition; Glycemic Variability
MeSH Terms: conditions — Critical Illness; Hyperglycemia; Diabetes Mellitus | interventions — Fructose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet 1 (Active Comparator): Low-carbohydrate Enteral Formula With Fructose
  Interventions: Dietary Supplement: Enteral Formula With Fructose
- Diet 2 (Active Comparator): Low-carbohydrate Enteral Formula Without Fructose
  Interventions: Dietary Supplement: Enteral Formula Without Fructose

INTERVENTIONS:
Dietary Supplement: Enteral Formula With Fructose — Low-carbohydrate Enteral Formula With Fructose
  Arms: Diet 1
Dietary Supplement: Enteral Formula Without Fructose — Low-carbohydrate Enteral Formula Without Fructose
  Arms: Diet 2

SUMMARY:
Hyperglycemia is a known risk factor for mortality in critically ill patients. Most of these patients receive enteral feeding. There is controversy about ideal carbohydrate composition of these diets. The aim of this study was to compare an enteral formula with the same proportion of carbohydrates with and without fructose on blood glucose levels.

DETAILED DESCRIPTION:
Randomized, cross-over, controlled, double-blind clinical trial without washout. Adult patients admitted to the ICU who presented capillary glycemia values> 180mg / dl with a full and exclusive enteral diet. They were randomized and observed for 4 days (2 days with each diet: with / without fructose). Capillary glycemia was measured 4 / 4h.

ELIGIBILITY:
Inclusion Criteria:

* Critical Illness
* Exclusive enteral diet
* Enteral diet with full nutritional value
* Hyperglycemia ≥180 mg / dl

Exclusion Criteria:

* Oral feeding
* NPT (Total or Partial Parenteral Nutrition)
* Patient without indication of use of study diets

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Glycemic Variability | four days
  To evaluate the glycemic oscillation during the use of enteral feedings

IPD SHARING:
Plan to Share IPD: No